CLINICAL TRIAL: NCT01252862
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on One Topical Hypotensive Medication Treated With Two Trabecular Micro-bypass Stents
Brief Title: Prospective Evaluation of Open-Angle Glaucoma Subjects on One Topical Hypotensive Medication Treated With Two iStents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-017
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Subjects With Primary Open-angle Glaucoma (POAG)
Keywords: Open angle; Glaucoma; Surgery; Ocular Hypertension; eye diseases
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two iStents devices (Experimental): Two iStents devices will be implanted
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent — Implantation of two iStents through a small temporal clear corneal incision

SUMMARY:
The purpose of this study is to evaluate the intraocular pressure (IOP) lowering effect of two iStent devices in eyes of subjects with primary open-angle glaucoma

DETAILED DESCRIPTION:
This study evaluates the safety and efficacy of two iStents implanted in primary open-angle glaucoma subjects

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subject on one topical hypotensive medication

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP reduction of greater than or equal to 20% at month 12 vs baseline | 12 Months

SECONDARY OUTCOMES:
IOP < 18 mm Hg at Month 12 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- S.V. Malayan's Ophthalmology Centre, Yerevan, Armenia

REFERENCES:
- [Background] Donnenfeld ED, Solomon KD, Voskanyan L, Chang DF, Samuelson TW, Ahmed II, Katz LJ. A prospective 3-year follow-up trial of implantation of two trabecular microbypass stents in open-angle glaucoma. Clin Ophthalmol. 2015 Nov 3;9:2057-65. doi: 10.2147/OPTH.S91732. eCollection 2015. PMID 26604675